CLINICAL TRIAL: NCT00083330
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Recombinant Multiclade HIV-1 Adenoviral Vector Vaccine, VRC-HIVADV014-00-VP, in Uninfected Adult Volunteers
Brief Title: Safety and Immunogenicity of an HIV Vaccine in Normal Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040172; 04-I-0172
Record Dates: First submitted 2004-05-20; First posted 2004-05-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-01

CONDITIONS: Healthy; HIV Infections
Keywords: Healthy; T Cells; Immunity; Healthy Volunteer; HV
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: VRC-HIVADV014-00-VP

SUMMARY:
This study will test the safety of an experimental vaccine against HIV infection and see if it causes an immune response to HIV. The vaccine is given by injection (shot) in the upper arm. It is made from DNA that codes for three HIV proteins. The DNA is inserted into an adenovirus that carries it into the muscle cells. The adenovirus normally can cause eye or upper respiratory infections, such as a cold; however, for the vaccine, it has been modified so that it cannot cause illness. Nor can the vaccine cause HIV infection, because it codes for only three of the nine HIV proteins.

Healthy, normal volunteers between 18 and 44 years of age who are not HIV-infected may be eligible for this study. Candidates are screened with a medical history and physical examination and blood and urine tests.

Participants are randomly assigned to receive either the experimental vaccine or a placebo (an inactive substance that looks like the vaccine). The vaccine or placebo is administered to participants in groups, according to their entry into the study. The first group receives the lowest study dose of vaccine. If this dose is safe, then the second group receives a higher dose. If this dose is also safe, then the third and final group receives the highest study dose. Clinic staff observe the subjects for side effects for 30 minutes after the injection, and subjects keep a diary card for the next 5 days, recording their temperature and any symptoms that may appear. Subjects are contacted by a nurse 2 days after the injection for follow-up.

Participants are seen at the clinic for follow-up visits 1, 2, 4, 12, and 24 weeks after the injection, and then are contacted by telephone for follow-up once a year until 5 years after the injection. The clinic visits include a physical examination, medical history, blood and urine tests, and HIV counseling, as needed. Women have pregnancy tests at the screening evaluation and again at study week 24. All subjects are tested for HIV at screening and at study weeks 12 and 24, and all subjects complete a "social impact questionnaire" at week 24. All subjects are asked questions about their sexual behavior and drug use.

...

DETAILED DESCRIPTION:
Study Design:

This is a Phase I, randomized, placebo-controlled, double-blinded study to examine safety, tolerability and immune response of a multiclade HIV adenoviral vector vaccine in uninfected adults. The hypothesis is that this vaccine will be safe and elicit immune responses to HIV. The primary objective is to evaluate the safety and tolerability of VRC-HIVADV014-00-VP in uninfected subjects and the secondary objectives include immunogenicity evaluations and adenovirus serotype 5 (Ad5) antibody titers through Week 4 and social impacts at Week 24. Exploratory evaluations include immunogenicity evaluations at Weeks 12 and 24 and Ad5 antibody titers at Week 24.

Product Description:

VRC-HIVADV014-00-VP is a recombinant product composed of 4 adenoviral vectors (Ad) (in a 3:1:1:1 ratio) that encode the HIV-1 Gag/Pol polyprotein from clade B and HIV-1 Env glycoproteins from clades A, B, and C, respectively. The final formulation buffer, VRC-DILUENT013-DIL-VP will be used as the diluent and as the placebo control. Injections will be administered intramuscularly (IM).

Subjects:

Healthy adult volunteers (18 to 44 years old).

Study Plan:

Thirty-six volunteers will receive one 1.0 mL injection of the study agent or placebo in a deltoid muscle as shown in the schema. Dose escalation will occur about three weeks after the last injection in a dose group following an interim safety data review by a DSMB, provided that there are no significant toxicities.

Study Duration:

Subjects will be evaluated at 5 or more clinical visits for 24 weeks after the study injection, followed by annual telephone or mail contact for the subsequent 4 years.

Study Endpoints:

The primary endpoint is safety of the vaccine administered at doses of 1 x 10(9), 1 x 10(10) and 1 x 10(11) particle units (PU) by intramuscular injection. Secondary endpoints are immunogenicity as indicated by HIV-specific antibody and cellular immune responses through Week 4, Ad5 antibody titer at Week 0 and Week 4 and social impact at Week 24. Exploratory analyses of immunogenicity at Weeks 12 and 24 and Ad5 antibody titer at Week 24 will also be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

18 to 44 years old.

Available for clinical follow-up through Week 24 and telephone or mail contact for an additional 4 years.

Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.

Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.

Able and willing to complete the informed consent process.

Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.

Willing to donate blood for sample storage to be used for future research.

Willing to discuss HIV infection risks and amenable to risk reduction counseling.

In good general health without clinically significant medical history.

Physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment.

Laboratory Criteria within 28 days prior to enrollment:

Hemoglobin is greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men

WBC is equal to 3,300-12,000 cells/mm(3)

Differential either within institutional normal range or accompanied by site physician approval

Total lymphocyte count is greater than or equal to 800 cells/mm(3)

Platelets is equal to 125,000 - 550,000/mm(3)

ALT (SGPT) is less than or equal to upper limit of normal

Serum creatinine is less than or equal to upper limit of normal

Normal urinalysis defined as negative glucose, negative or trace protein, and negative or trace hemoglobin (blood).

Negative FDA-approved HIV blood test

Negative Hepatitis B surface antigen

Negative anti-HCV

Female-Specific Criteria:

Negative Beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential.

A female participant must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation.,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 24 of the study,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 24 of the study by one of the following methods:

* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply.

Women:

Breast-feeding.

Volunteer has received any of the following substances:

HIV vaccines in a prior clinical trial

Immunosuppressive or cytotoxic medications within the past six months with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis

Blood products within 120 days prior to HIV screening

Immunoglobulin within 60 days prior to HIV screening

Live attenuated vaccines within 30 days prior to initial study vaccine administration

Investigational research agents within 30 days prior to initial study vaccine administration

Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration

Current anti-TB prophylaxis or therapy

Volunteer has a history of any of the following clinically significant conditions:

Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain

Autoimmune disease or immunodeficiency

Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.

Diabetes mellitus (type I or II), with the exception of gestational diabetes.

History of thyroidectomy or thyroid disease that required medication within the past 12 months.

Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.

Blood pressure that is more than 145/95 at enrollment or hypertension that requires medication.

Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.

Syphilis infection that is active or a positive serology due to a syphilis infection treated less than six months ago.

Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.

Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.

Asplenia or any condition resulting in the absence or removal of the spleen.

Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.

Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36
Dates: Start 2004-05-18; Primary Completion 2009-10-01 (Actual); Study Completion 2009-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Borrow P, Lewicki H, Hahn BH, Shaw GM, Oldstone MB. Virus-specific CD8+ cytotoxic T-lymphocyte activity associated with control of viremia in primary human immunodeficiency virus type 1 infection. J Virol. 1994 Sep;68(9):6103-10. doi: 10.1128/JVI.68.9.6103-6110.1994. PMID 8057491
- [Background] Koup RA, Safrit JT, Cao Y, Andrews CA, McLeod G, Borkowsky W, Farthing C, Ho DD. Temporal association of cellular immune responses with the initial control of viremia in primary human immunodeficiency virus type 1 syndrome. J Virol. 1994 Jul;68(7):4650-5. doi: 10.1128/JVI.68.7.4650-4655.1994. PMID 8207839
- [Background] Pantaleo G, Demarest JF, Soudeyns H, Graziosi C, Denis F, Adelsberger JW, Borrow P, Saag MS, Shaw GM, Sekaly RP, et al. Major expansion of CD8+ T cells with a predominant V beta usage during the primary immune response to HIV. Nature. 1994 Aug 11;370(6489):463-7. doi: 10.1038/370463a0. PMID 8047166
- [Derived] Catanzaro AT, Koup RA, Roederer M, Bailer RT, Enama ME, Moodie Z, Gu L, Martin JE, Novik L, Chakrabarti BK, Butman BT, Gall JG, King CR, Andrews CA, Sheets R, Gomez PL, Mascola JR, Nabel GJ, Graham BS; Vaccine Research Center 006 Study Team. Phase 1 safety and immunogenicity evaluation of a multiclade HIV-1 candidate vaccine delivered by a replication-defective recombinant adenovirus vector. J Infect Dis. 2006 Dec 15;194(12):1638-49. doi: 10.1086/509258. Epub 2006 Nov 8. PMID 17109335